CLINICAL TRIAL: NCT06334627
Title: Every Newborn-Reach Up Early Education Intervention for All Children- a Parent Group Intervention for School Readiness in Bangladesh, Nepal, and Tanzania
Acronym: EN-REACH
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: International Centre for Diarrhoeal Disease Research, Bangladesh (Other); Golden Community, Nepal (Unknown); Muhimbili University of Health and Allied Sciences (Other); University of Glasgow (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Supportive Care
Other Study IDs: ENREACH
Record Dates: First submitted 2024-02-29; First posted 2024-03-28 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-02

CONDITIONS: Child Development; Child Development Disorder
Keywords: Child development; child disability; pre-primary education; school readiness
MeSH Terms: conditions — Developmental Disabilities

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-Primary Intervention (Experimental): Program consisting of 9 modules focussing on early learning, play, saftey, wellbeing, reading and writing will be delivered approximately every two weeks to groups of 10 parents from the intervention arm.
  Interventions: Behavioral: Pre-Primary Intervention
- Control (No Intervention): No intervention delivered. Participants will attend any government pre-primary based programmes as standard of care.

INTERVENTIONS:
Behavioral: Pre-Primary Intervention — School readiness intervention
  Arms: Pre-Primary Intervention

SUMMARY:
The goal of this clinical trial is to test the effect of a pre-primary education parent group intervention in children with and without disability in Nepal Bangladesh and Tanzania. The main question it aims to answer are:

* What is the impact of a parent group intervention on primary school readiness in children aged 5-6 years old in three LMICs?
* What is the feasibility and accessibility of a parent group intervention for these children?

Participants will attend parent group sessions every two weeks for a total of 9 sessions. Researchers will compare a control group to see if there are impacts on school readiness and child development.

DETAILED DESCRIPTION:
Vulnerable children, including those with neuro-developmental delays and disabilities, often face barriers in accessing early primary education, thus hindering progress toward Sustainable Development Goal 4.2. Evidence-based interventions are essential to enhancing inclusivity and establishing sustainable implementation strategies to address this challenge. This study, Every Newborn - Reach up Early Education Intervention for All Children (EN-REACH), builds on the previous Every Newborn- Simplified Measurement Integrating Longitudinal Neurodevelopmental and Growth (EN-SMILING) observational cohort study. This is a cluster randomized controlled trial (cRCT) to evaluate the effectiveness of a parenting group intervention program for enhancing school readiness in Bangladesh, Nepal, and Tanzania, and an embedded process evaluation to inform scalability and feasibility.

EN-REACH is a cRCT with 150 clusters to evaluate the impact of a parent training program led by trained parent-teacher facilitator pairs, focusing on children aged 4~6 years preparing for preschool. Approximately 500 participants from the EN-SMILING cohort at each site have been identified. A geographic information system will define ~50 clusters in each of the three countries, each with approximately ten parent-child dyads. Half the clusters will be randomly assigned to intervention and control groups. The primary outcome is "school readiness", assessed using the Measuring Early Learning Quality and Outcomes (MELQO) tool. Secondary outcomes include Intelligence Quotient, child functioning, growth, visual, and hearing assessments. Data will be collected at baseline, and post-intervention data following implementation of the parent group intervention sessions over approximately 5-months. Quantitative data on coverage and quality care, combined with qualitative insights from children, caregivers, facilitators, and stakeholders' perspectives, will be used to conduct a process evaluation applying the RE-AIM framework.

This trial focused on enhancing school readiness and cognitive abilities in young children, inclusive of those with disabilities, aims to bridge gap from home to early primary education. EN-REACH aims to provide insights into the effectiveness and acceptability of a co-designed disability-inclusive school readiness program in three countries, potentially impacting national, and global policies for all children, including those with disabilities.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 4-6 years in study area
* Children who completed previous EN-SMILING Study

Exclusion Criteria:

* Children outside of age range
* Children living outside of study area

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1651 (Actual)
Dates: Start 2022-05-03 (Actual); Primary Completion 2024-04-15 (Estimated); Study Completion 2024-09-15 (Estimated)

PRIMARY OUTCOMES:
Measuring Early Learning Quality and Outcomes (MELQO Tool) | Baseline (children are aged 5-5.5 years) and 6 months later post intervention (children aged 5.5-6 years)
  School Readiness
The Pediatric Evaluation of Disability Inventory | Baseline (children are aged 5-5.5 years) and 6 months later post intervention (children aged 5.5-6 years)
  Child Disability

SECONDARY OUTCOMES:
Washington Group Questionnaire | Baseline (children are aged 5-5.5 years) and 6 months later post intervention (children aged 5.5-6 years)
  Child functioning
The Wechsler Preschool & Primary Scale of Intelligence | Baseline (children are aged 5-5.5 years) and 6 months later post intervention (children aged 5.5-6 years)
  Child IQ
Pre-school Register | Baseline (children are aged 5-5.5 years) and 6 months later post intervention (children aged 5.5-6 years)
  Pre-school attendance
Mental Health Questionnaire | Baseline (children are aged 5-5.5 years) and 6 months later post intervention (children aged 5.5-6 years)
  Maternal Mental Health screen
Pediatric Quality of Life Inventory (PEDSQL Tool) | Baseline (children are aged 5-5.5 years) and 6 months later post intervention (children aged 5.5-6 years)
  Child and family quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Joy Lawn, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (3):
- International Centre for Diarrheal Disease Research, Bangladesh, Dhaka, Bangladesh
- Golden Community, Lalitpur, Nepal
- Muhimbili University of Health and Allied Sciences, Dar es Salaam, Tanzania

IPD SHARING:
Plan to Share IPD: Undecided
Annonomysed primary outcome data will be made available along with the protocol and statistical analysis plan

REFERENCES:
- [Derived] Miah MAA, Chandna J, Gurung R, Masoud NS, Paul P, Ameen S, Basnet O, Miraji M, Tann C, Mili IA, Hossain AKMT, Chowdhury AI, Alam A, Milner KM, Arifeen SE, Kc A, Manji K, Lynch P, Lawn JE, Hamadani JD; EN-REACH collaborative group. Every Newborn-Reach Up Early Education Intervention for All Children (EN-REACH)- a parent group intervention for school readiness in Bangladesh, Nepal, and Tanzania: study protocol for a cluster randomized controlled trial. Trials. 2024 Aug 23;25(1):556. doi: 10.1186/s13063-024-08381-6. PMID 39180108